CLINICAL TRIAL: NCT01012336
Title: Safety and Efficacy of Aprepitant, Ramosetron, and Dexamethasone for Chemotherapy-Induced Nausea and Vomiting in Patients With Ovarian Cancer Treated With Taxane/Carboplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-09-119
Record Dates: First submitted 2009-11-10; First posted 2009-11-13 (Estimated); Results first posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-10

CONDITIONS: Chemotherapy-Induced Nausea and Vomiting; Ovarian Cancer
Keywords: efficacy and safety of Aprepitant/Ramosetron/Dexamethasone in ovary cancer patients with taxol and carboplatin
MeSH Terms: conditions — Vomiting; Ovarian Neoplasms | interventions — Aprepitant

ARMS (1):
- Aprepitant (Experimental)
  Interventions: Drug: Aprepitant/Ramosetron/Dexamethasone

INTERVENTIONS:
Drug: Aprepitant/Ramosetron/Dexamethasone — Aprepitant: The first day, one 125 mg capsule will be administered per oral, 1 hour before chemotherapy. Thereafter one 80 mg capsule will be repeated daily between 8 to 10 a.m. during days 2 to 3.
  Ramosetron: 0.3 mg i.v. a single dose on day 1, administered over 30 seconds, 30 minutes prior to chemotherapy.
  Dexamethasone: 20mg diluted in 50ml of 0.9% saline i.v. a single dose on day 1, administered over 30minutes prior to chemotherapy (taxane). Because all patients are premedicated with dexamethasone 20 mg before taxane administration, the dose of dexamethasone can not be reduced to 12 mg.

SUMMARY:
The current recommended guideline for patients receiving moderately emetogenic chemotherapy (MEC) is the combination of a 5-HT3 receptor antagonist and corticosteroid. Incidence of chemotherapy induced nausea and vomiting (CINV) is approximately 50% in patients receiving MEC. An incidence rate of 25-38% for delayed emesis and 55-60% for delayed nausea has been observed. Hence, there is clearly a need for more effective prevention of CINV in patients receiving MEC, especially in women with ovarian carcinoma who are particularly susceptible to these symptoms. Therefore the investigators designed a study with the objective to evaluate if new combination (Aprepitant/Ramosetron/Dexamethasone) may improve actual CINV control in ovarian carcinoma patients treated with taxane/carboplatin.

ELIGIBILITY:
Inclusion criteria

1. patient is over 18 years
2. ovarian carcinoma patients who are treated with moderately emetogenic chemotherapy
3. Karnofsky score > 60
4. Life expectancy > 4 months

Exclusion criteria

1. Any of following conditions (mentally incapacitated or emotional or psychiatric disorder, user of any illicit drugs, has an active infection, hypersensitivity to ramosetron or aprepitant)
2. Patients have received a nonapproved drug within last 4 weeks
3. abnormal laboratory values (AST > 2.5 normal, ALT > 2.5 normal, Bilirubin > 1.5 normal, Creatinine > 1.5 normal)
4. Antiemetic drugs within 48 hours of study
5. Benzodiazepine or opiate within 48 hours
6. CYP3A4 substrates within 7 days (terfenadine, cisapride, astemizole, pimozide)
7. CYP3A4 inhibitors (clarithromycin, ketoconazole)
8. CYP3A4 inducers within 30 days (Barbiturates, rifampicin, carbamazepine)

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duk Soo Bae, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Choi CH, Kim MK, Park JY, Yoon A, Kim HJ, Lee YY, Kim TJ, Lee JW, Kim BG, Bae DS. Safety and efficacy of aprepitant, ramosetron, and dexamethasone for chemotherapy-induced nausea and vomiting in patients with ovarian cancer treated with paclitaxel/carboplatin. Support Care Cancer. 2014 May;22(5):1181-7. doi: 10.1007/s00520-013-2070-6. Epub 2013 Dec 12. PMID 24337621

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant: Aprepitant is a selective, high-affinity NK1 receptor antagonist. Patients received the following regimen (Day 1: aprepitant 125 mg, ramosetron 0.6 mg, and dexamethasone 20 mg before chemotherapy; Days 2-3: aprepitant 80 mg every day)
Period: Overall Study
Arm/Group | Aprepitant
Started | 85
Completed | 85
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Aprepitant: Aprepitant is a selective, high-affinity NK1 receptor antagonist
Arm/Group | Aprepitant
Number analyzed (Participants) | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 69
  >=65 years | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 54.9 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85
  Male | 0
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 85

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of the Aprepitant/Ramosetron/Dexamethasone Regimen in Terms of the Proportion of Patients With a Complete Response (CR) During the 120 Hour Following Initiation of Chemotherapy.
Description: Complete Response is defined as No vomiting with no rescue therapy. These response criteria will be applied to the following time periods: Overall: from 0 (chemotherapy initiation) to the morning of day 6, Acute: 0 to 24 hours following the initiation of chemotherapy, Delayed: 25 hours to the morning of day 6(D6).
Time Frame: 120 hours
Measure: Number; unit: Percentage of Participants
Groups:
- Aprepitant: Aprepitant is a selective, high-affinity NK1 receptor antagonist. Patients received the following regimen (Day 1: aprepitant 125 mg, ramosetron 0.6 mg, and dexamethasone 20 mg before chemotherapy; Days 2-3: aprepitant 80 mg every day)
Arm/Group | Aprepitant
Number analyzed (Participants) | 85
Percentage of Participants | 89.4

2. Primary Outcome: Safety and Tolerability of the Aprepitant/Ramosetron/Dexamethasone Regimen
Time Frame: 120 hours
Reporting Status: Not Posted

3. Secondary Outcome: Efficacy of the Aprepitant/Ramosetron/Dexamethasone Regimen in Terms of the Proportion of Patients With no Vomiting During the 120 Hour Following Initiation of Chemotherapy
Time Frame: 120 hours
Reporting Status: Not Posted

4. Secondary Outcome: Time to First Vomiting Episode or Use of Rescue Medication
Time Frame: 120 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Aprepitant
Serious Adverse Events (participants affected / at risk) | 2/89
Other Adverse Events (participants affected / at risk) | 35/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant (N=89)
Neutropenic fever (Blood and lymphatic system disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant (N=89)
constipation (Gastrointestinal disorders) | 14 (14)
fatigue (General disorders) | 13 (13)
headache (Nervous system disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes